CLINICAL TRIAL: NCT06912412
Title: Development and Validation of a Community-Based Remote Cardiac Rehabilitation Program for Improving Cardiopulmonary Function and Quality of Life in Pediatric Patients With Complex Congenital Heart Disease
Brief Title: Community-Based Remote Cardiac Rehabilitation Program for Pediatric Patients With Complex Congenital Heart Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: University of Seoul (Other)
Responsible Party: Principal Investigator, Woo Hyung Lee, Clinical associate professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FP-2024-00016
Record Dates: First submitted 2025-03-16; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Congenital Heart Disease (CHD); Complex Congenital Heart Disease; Congenital Heart Disease in Children
Keywords: Complex congenital heart disease; remote cardiac rehabilitation; cardiac rehabilitation; children cardiac rehabilitation
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Community-based remote cardiac rehabilitation group (Experimental): The group is provided with a single session of supervised remote cardiac rehabilitation session per week, and 4 sessions of home-based rehabilitation.
  During the supervised remote session, the EKG signal, heart rate and SpO2 of the participants are monitored in real-time using a single lead EKG and SpO2 monitor. Their activity levels are also recorded using a smartwatch, in number of steps and minutes in moderate-vigorous physical activity time
  Interventions: Other: Community-based supervised remote cardiac rehabilitation; Other: Home-based cardiac rehabilitation program

INTERVENTIONS:
Other: Community-based supervised remote cardiac rehabilitation — Community-based supervised remote cardiac rehabilitation begins with a weekly session led by exercise specialists, who use remote-based materials to match each participant's target heart rate and rate of perceived exertion (RPE). During these sessions, participants perform aerobic, strength, and respiratory exercises using progressive overload principles, with devices such as the POWERbreathe Plus supporting individualized respiratory training.
  Depending on the risk classification for each participant, they will be provided with different intensity of exercises (depending on their measured HR max, HRR, and/or RPE).
Other: Home-based cardiac rehabilitation program — Beyond the single supervised session, participants undertake four weekly home-based sessions.
  * Low-Risk Group: Aerobic and respiratory exercises are performed four times per week, plus strength training once or twice weekly. Each 60-minute session includes a 10-minute warm-up, 40-minute main exercise, and 10-minute cool-down. Indoor sessions use remote exercise content and respiratory training devices, while outdoor activities may involve walking, jogging, cycling, or swimming. Exercises progress in duration, intensity, and resistance.
  * Moderate-Risk Group: Aerobic and respiratory exercises are done four times per week with an RPE of 8-13. Intensity and duration increase gradually, contingent on symptom stability and improved endurance.
  * High-Risk Group: Aerobic and respiratory sessions occur four times a week at an RPE of 8-10, each lasting around 30 minutes (5-minute warm-up, 20-30-minute main exercise, 5-minute cool-down).

SUMMARY:
This study is to develop a 12-week community-based remote cardiac rehabilitation program for pediatric patients with complex congenital heart disease and to assess its validity and safety.

For these children, a multidisciplinary approach including pediatric rehabilitation medicine, pediatric thoracic surgery, pediatrics, pediatric psychiatry, sports science, and nutrition is essential, but such comprehensive services are rarely available in Korea. As a result, pediatric cardiac rehabilitation at the community level is nearly nonexistent. Recent long-term retrospective cohort studies suggest that maintaining regular physical activity and aerobic capacity from early childhood significantly reduces future cardiovascular complications, emphasizing the importance of early pediatric cardiac rehabilitation. However, participation in existing programs is low due to limited accessibility.

The investigators hypothesize that a community-based remote cardiac rehabilitation program for these patients is both valid and safe. Participants will be children aged 8-18 years diagnosed with complex congenital heart disease , at least 3 months post-surgery, and stable cardiovascular status.

Interventions include supervised and self-directed cardiac rehabilitation exercises. Monitoring (heart rate, SpO2, ECG) will be performed in real-time, with non-real-time data collection of physical activity using smartwatches. The intervention lasts 12 weeks with a 12-week follow-up.

Validity measures include baseline evaluation, adherence, dropout rate, participant and parent satisfaction, and changes in cardiopulmonary exercise capacity, physical activity, body composition, fitness (6-minute walk, strength, flexibility, respiratory muscle strength), and questionnaires (physical activity, quality of life, exercise satisfaction, depression, psychological state).

Safety will be assessed by monitoring adverse events, vital signs, fatigue (Borg scale), and pain before and after exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 8 and 18 years
2. Diagnosed with complex congenital heart disease (Complex CHD) and have undergone surgery
3. At least 3 months post-cardiac surgery with a stable hemodynamic status
4. Capable of using remote programs (e.g., mobile apps, video-conferencing platforms) at home, with technical support from a caregiver
5. Either the participant or their caregiver agrees to study participation and has signed the informed consent form

Exclusion Criteria:

1. Patients with uncontrolled arrhythmias, acute heart failure, myocarditis, pericarditis, or other ongoing cardiovascular conditions.
2. Patients who are unable to exercise independently due to neurological or musculoskeletal disorders.
3. Patients who cannot understand or carry out remote rehabilitation program instructions due to cognitive impairment.
4. Patients showing clinically significant levels of depression or anxiety on the CDI-2 or RCMAS.
5. Patients who cannot cooperate with required study assessments (e.g., CPET, ECG, 6MWT).

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Drop-out rate | baseline, 12 weeks after, 24 weeks after follow-up
Attendance rate | baseline, 12 weeks after, 24 weeks after follow-up

SECONDARY OUTCOMES:
oxygen consumption, VO2 | baseline, 12 weeks after, 24 weeks after follow-up
  Oxygen consumption (VO2) refers to the rate at which the body takes in and uses oxygen.
maximal oxygen consumption, VO2 max | baseline, 12 weeks after, 24 weeks after follow-up
  Maximal oxygen consumption (VO2 max) represents the highest rate at which an individual can take in, transport, and utilize oxygen during maximal or exhaustive exercise.
Respiratory exchange rate, RER | baseline, 12 weeks after, 24 weeks after follow-up
  Respiratory Exchange Ratio (RER) is the ratio of the volume of carbon dioxide produced (VCO2) to the volume of oxygen consumed (VO2) in the body.
  RER = VCO2 / VO2
minute ventilation (VE) | baseline, 12 weeks after, 24 weeks after follow-up
  minute ventilation (VE) refers to the total volume of air inhaled or exhaled by an individual per minute.
  VE = Tidal Volume (VT) x Respiratory Rate (RR)
ventilation effectiveness, VE/VO2 | baseline, 12 weeks after, 24 weeks after follow-up
  Ventilation effectiveness, when expressed as the ratio of minute ventilation (VE) to oxygen consumption (VO2) (VE/VO2), represents the volume of air that needs to be breathed to consume one liter of oxygen.
oxygen per pulse, O2 pulse | baseline, 12 weeks after, 24 weeks after follow-up
oxygen saturation, SpO2 | baseline, 12 weeks after, 24 weeks after follow-up
maximal heart rate during exercise, HR max | baseline, 12 weeks after, 24 weeks after follow-up
heart rate by exercise intensity | baseline, 12 weeks after, 24 weeks after follow-up
average number of steps for 7 days using smartwatch | baseline, 12 weeks after, 24 weeks after follow-up
average moderate-vigorous physical activity time for 7days using smartwatch, minutes | baseline, 12 weeks after, 24 weeks after follow-up
skeletal muscle mass (kg) | baseline, 12 weeks after, 24 weeks after follow-up
body fat mass (kg) | baseline, 12 weeks after, 24 weeks after follow-up
body fat percentage | baseline, 12 weeks after, 24 weeks after follow-up
Abdominal fat percentage | baseline, 12 weeks after, 24 weeks after follow-up
Intracellular moisture, extracellular moisture | baseline, 12 weeks after, 24 weeks after follow-up
Radial artery pulse wave amplification index: Augmentation index (AIx@75 index) | baseline, 12 weeks after, 24 weeks after follow-up
  arterial stiffness and wave reflection at a heart rate of 75 beats per minute
Carotid-femoral pulse wave velocity, c-f PWV | baseline, 12 weeks after, 24 weeks after follow-up
  Carotid-femoral pulse wave velocity (c-f PWV) is a non-invasive medical test used to assess arterial stiffness, which is a measure of how rigid or flexible the arteries are.
  c-f PWV = Distance between carotid and femoral sites / Time difference between pulse wave arrival at the two sites.
Flow-mediated dilation, FMD% | baseline, 12 weeks after, 24 weeks after follow-up
  Flow-Mediated Dilation (FMD%) is a non-invasive ultrasound technique used to assess endothelial function, which is the ability of the inner lining of arteries (the endothelium) to relax and contract properly. FMD% specifically measures the percentage change in the diameter of an artery in response to an increase in blood flow
6 minutes walk test | baseline, 12 weeks after, 24 weeks after follow-up
  total distance in meters
lower limb muscle strength test (peak torque/BW) | baseline, 12 weeks after, 24 weeks after follow-up
Upper extremity strength test: grip force (kg) | baseline, 12 weeks after, 24 weeks after follow-up
Flexibility check: Flexibility distance (cm) | baseline, 12 weeks after, 24 weeks after follow-up
Respiratory muscle strength test (MIP mmH2O) | baseline, 12 weeks after, 24 weeks after follow-up
  Maximal Inspiratory Pressure (MIP) is a measurement in assessing the strength of inspiratory muscles. It reflects the strength of the diaphragm and other inspiratory muscles.
Global Physical Activity Questionnaire | baseline, 12 weeks after, 24 weeks after follow-up
  The Global Physical Activity Questionnaire (GPAQ) doesn't have a fixed minimum and maximum score.
  A score of 0 would indicate no reported physical activity. Higher scores means a better outcome in terms of physical activity levels.
Pediatric Quality of Life Inventory™ (PedsQL™) for subjects and parents | baseline, 12 weeks after, 24 weeks after follow-up
  Minimum Value (Total Score): 0 Maximum Value (Total Score): 100 Higher Scores Mean: A better outcome. Higher scores on the PedsQL™ indicate a better health-related quality of life, as reported by either the child/adolescent or their parent.
Pediatric Quality of Life Inventory Cardiac, PedsQL™ Cardiac | baseline, 12 weeks after, 24 weeks after follow-up
  Minimum Value (Total Score): 0 Maximum Value (Total Score): 100 Higher Scores Mean: A better outcome. Higher scores on the PedsQL™ Cardiac module indicate a better health-related quality of life for the child with a cardiac condition.
Program satisfactory survey | 12 weeks
Resilience Scale for Youth, RS-Y | baseline, 12 weeks after, 24 weeks after follow-up
  Minimum Value: 25 Maximum Value: 125 Higher Scores Mean: A better outcome. Higher scores on the Resilience Scale for Youth indicate a higher level of resilience in the individual.
Child Behavior Checklist for parents, CBCL | baseline, 12 weeks after, 24 weeks after follow-up
  Minimum Value : 0 Maximum Value : 118 Higher Scores Mean: A worse outcome. Higher scores on the Total Problems scale of the CBCL indicate a greater number and severity of reported behavioral and emotional problems in the child.
blood pressure by exercise intensity | baseline, 12 weeks after, 24 weeks after follow-up
Children's Depression Inventory 2, K-CDI-2:SR | baseline, 12 weeks after, 24 weeks after follow-up
  Minimum Value: 0 Maximum Value: 54 Higher Scores Mean: A worse outcome. Higher scores on the K-CDI-2:SR indicate higher levels of reported depressive symptoms.
Revised Children's Manifest Anxiety Scale 2, RCMAS-2 | baseline, 12 weeks after, 24 weeks after follow-up
  Minimum Value: 0 Maximum Value: 49 Higher Scores Mean: A worse outcome. Higher scores on the RCMAS-2 indicate higher levels of reported anxiety.
Incidence proportion of adverse events and harm during exercise | 12 weeks after, 24 weeks after follow-up
  Incidence proportion of participants with exercise-related adverse events as assessed by CTCAE v4.0
Incidence rate of adverse events and harm during exercise | 12 weeks after, 24 weeks after follow-up
  Incidence rate of participants with exercise-related adverse events as assessed by CTCAE v4.0
Changes in pre- and post-workout heart rate | up to 12 weeks
Changes in pre- and post-workout oxygen saturation (SpO2) | up to 12 weeks
Changes in pre- and post-workout respiratory rate | up to 12 weeks
Rate of Perceived Exertion, Borg scale | up to 12 weeks
  Unabbreviated Scale Title: Rate of Perceived Exertion (RPE) Scale Minimum Value: 6 Maximum Value: 20 Higher Scores Mean: A worse outcome. Higher numbers on the Borg scale indicate a greater feeling of exertion.
Upper extremity strength test: relative grip force (%) | baseline, 12 weeks after, 24 weeks after follow-up
lower limb muscle strength test (peak torque) | baseline, 12 weeks after, 24 weeks after follow-up
extracellular moisture ratio | baseline, 12 weeks after, 24 weeks after follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided